CLINICAL TRIAL: NCT05555329
Title: Alternative Dosing Scheme of Pomalidomide 4 mg Every Other Day Versus Pomalidomide 2 mg and 4 mg Every Day: Reduction in Costs, Same Efficacy? A PKPD Bioequivalence Pilot Study; the POMAlternative Study
Brief Title: Alternative Dosing Scheme of Pomalidomide 4 mg Every Other Day Versus Pomalidomide 2 mg and 4 mg Every Day; the POMAlternative Study
Acronym: POMAlternative
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Sonja Zweegman, MD, PhD, Professor of Hematology, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: POMAlternative
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma; Multiple Myeloma, Refractory
Keywords: Multiple myeloma; Pomalidomide; Pharmacokinetics/dynamics; Cost-effectiveness
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A; Pomalidomide 4 mg every other day in cycle 2 (Experimental): Group A (6 patients): Cycle 1: Pomalidomide 4 mg every day on day 1-21; Cycle 2: 4 mg every other day on day 1-21; Cycle 3: 2 mg every day on day 1-28. In Cycles of 28 days.
  Interventions: Drug: Pomalidomide 4 mg every day in cycle 1; Drug: Pomalidomide 4 mg every other day in cycle 2; Drug: Pomalidomide 2 mg every day in cycle 3
- Group B; Pomalidomide 4 mg every other day in cycle 3 (Experimental): Group B (6 patients): Cycle 1: Pomalidomide 4 mg every day on day 1-21; Cycle 2: 2 mg every day on day 1-28; Cycle 3: 4 mg every other day on day 1-21. In Cycles of 28 days.
  Interventions: Drug: Pomalidomide 4 mg every day in cycle 1; Drug: Pomalidomide 2 mg every day in cycle 2; Drug: Pomalidomide 4 mg every other day in cycle 3

INTERVENTIONS:
Drug: Pomalidomide 4 mg every day in cycle 1 — Pomalidomide 4 mg every day, on days 1-21 in a cycle of 28 days
  Other Names: Cycle 1
Drug: Pomalidomide 4 mg every other day in cycle 2 — Pomalidomide 4 mg every other day, on days 1-21 in a cycle of 28 days
  Other Names: Cycle 2 (Group A)
  Arms: Group A; Pomalidomide 4 mg every other day in cycle 2
Drug: Pomalidomide 2 mg every day in cycle 2 — Pomalidomide 2 mg every day, on days 1-28 in a cycle of 28 days
  Other Names: Cycle 2 (Group B)
  Arms: Group B; Pomalidomide 4 mg every other day in cycle 3
Drug: Pomalidomide 2 mg every day in cycle 3 — Pomalidomide 2 mg every day, on days 1-28 in a cycle of 28 days
  Other Names: Cycle 3 (Group A)
  Arms: Group A; Pomalidomide 4 mg every other day in cycle 2
Drug: Pomalidomide 4 mg every other day in cycle 3 — Pomalidomide 4 mg every other day, on days 1-21 in a cycle of 28 days
  Other Names: Cycle 3 (Group B)
  Arms: Group B; Pomalidomide 4 mg every other day in cycle 3

SUMMARY:
Pomalidomide either as single therapy or in combination with cyclophosphamide, elotuzumab, bortezomib, or daratumumab are effective treatment regimens in relapsed refractory multiple myeloma (RRMM). Standard dosing is 4 mg/day during 21 days of a 28-day cycle (21/28). However, a clear dose-response association for pomalidomide in patients with multiple myeloma (MM) is lacking. There is data supporting that a dose of 2 mg/day continuously (28/28) induces fewer side effects while efficacy is preserved, compared to 4 mg/day continuously. The response in patients who received pomalidomide 2 mg per day compared to 4 mg per day was higher, with a longer duration of response. In addition, a randomized phase II study showed no difference in efficacy between 4 mg (21/28) and 4 mg continuously. These clinical studies support that a dosage of pomalidomide of 2 mg (28/28) is at least comparable with a dosage of 4 mg (21/28). It is not known if 4 mg every other day (EOD) is comparable to a dosage of pomalidomide 2 mg (28/28) or 4 mg every day (QD, 21/28). For cost reasons, this is interesting as the costs of pomalidomide 4 mg and 2 mg are comparable. Therefore, from a patient and societal perspective, the investigators want to explore if an alternative scheme would be possible by performing a PKPD bio-equivalence pilot study.

DETAILED DESCRIPTION:
Pomalidomide either as single therapy or in combination with cyclophosphamide, elotuzumab, bortezomib, or daratumumab are effective treatment regimens in relapsed refractory multiple myeloma (RRMM). Standard dosing is 4 mg/day during 21 days of a 28-day cycle (21/28). However, a clear dose-response association for pomalidomide in patients with multiple myeloma (MM) is lacking. There is data supporting that a dose of 2 mg/day continuously (28/28) induces fewer side effects while efficacy is preserved, compared to 4 mg/day continuously. The response in patients who received pomalidomide 2 mg per day compared to 4 mg per day was higher, with a longer duration of response. In addition, a randomized phase II study showed no difference in efficacy between 4 mg (21/28) and 4 mg continuously. These clinical studies support that a dosage of pomalidomide of 2 mg (28/28) is at least comparable with a dosage of 4 mg (21/28). It is not known if 4 mg every other day (EOD) is comparable to a dosage of pomalidomide 2 mg (28/28) or 4 mg every day (QD, 21/28). For cost reasons, this is interesting as the costs of pomalidomide 4 mg and 2 mg are comparable. Therefore, from a patient and societal perspective, the investigators want to explore if an alternative scheme would be possible by performing a PKPD bio-equivalence pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory multiple myeloma, who are eligible for a treatment regimen which contains pomalidomide. Either monotherapy or in combination with bortezomib, daratumumab, cyclophosphamide, or elotuzumab
* Patients who received a minimum of two cycles of pomalidomide 4mg every day on day 1-21/28
* Age > 18 years
* WHO performance status 0-3
* Written informed consent

Exclusion Criteria:

* Usage of CYP1A2 inhibitors (e.g. ciprofloxacin, enoxacin, ketoconazole, carbamazepine, fluvoxamine, and grapefruit juice)
* Renal insufficiency requiring dialysis
* Significant hepatic dysfunction (total bilirubin > 330 μmol/l or transaminases > 3 times normal level)
* Current smoker
* Hemoglobin <6.5 mmol/L
* Thrombocytes <100 *10^9/L
* Neutrophiles <1.5 *10^9/L
* Pregnant patients
* Female patients who are able to get pregnant and who do not agree to adequate birth control or complete abstinence
* Male patients who do not agree to adequate birth control or complete abstinence
* Hypersensitivity to pomalidomide or constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
The AUC/MIC ratio | During three cycles of 28 days
  The AUC/MIC ratio during usage of pomalidomide 4 mg QD on day 1-21, 4 mg EOD on day 1-21, and 2 mg QD on day 1-28 in cycles of 28 days.
The level of the Ctrough | During three cycles of 28 days
  The level of the Ctrough during usage of pomalidomide 4 mg QD on day 1-21, 4 mg EOD on day 1-21, and 2 mg QD on day 1-28 in cycles of 28 days.

SECONDARY OUTCOMES:
Cmax | During three cycles of 28 days
  The Cmax during usage of pomalidomide 4 mg QD on day 1-21, 4 mg EOD on day 1- 21, and 2 mg QD on day 1-28 in cycles of 28 days.
Time above EC50 | During three cycles of 28 days
  The time above the EC50 during usage of pomalidomide 4 mg QD on day 1-21, 4 mg EOD on day 1- 21, and 2 mg QD on day 1-28 in cycles of 28 days.
Toxicity and side effects | During three cycles of 28 days
  Toxicity and side effects during usage of pomalidomide 4 mg every day on day 1-21, pomalidomide 4 mg every other day on day 1-21, and pomalidomide 2 mg every day on day 1-28 in cycles of 28 days.
Overall response rate (ORR) | During three cycles of 28 days
  Overall response rate (ORR), based on the IMWG criteria

OTHER OUTCOMES:
Explorative endpoint: T-cell activation | During three cycles of 28 days
  T-cell activation, defined as the expression of membrane activation markers and cytokine markers during usage of pomalidomide 4 mg every day on day 1-21, pomalidomide 4 mg every other day on day 1-21, and pomalidomide 2 mg every day on day 1-28 in cycles of 28 days.
Explorative endpoint: Ikaros/Aiolos degradation | During three cycles of 28 days
  Ikaros/Aiolos degradation as a biological measurement of pomalidomide activation during usage of pomalidomide 4 mg every day on day 1-21, pomalidomide 4 mg every other day on day 1-21, and pomalidomide 2 mg every day on day 1-28 in cycles of 28 days.
Explorative endpoint: Concentration of pomalidomide in PBMCs | During three cycles of 28 days
  Concentration of pomalidomide in PBMCs during usage of pomalidomide 4 mg every day on day 1-21, pomalidomide 4 mg every other day on day 1-21, and pomalidomide 2 mg every day on day 1-28 in cycles of 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Zweegman, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VUMedicalCenter, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No